CLINICAL TRIAL: NCT02250521
Title: McGRATH MAC Video Laryngoscope - To View or Not To View?
Brief Title: McGRATH MAC Video Laryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-14-0365
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-10

CONDITIONS: Intubation; Difficult
Keywords: BMI < 50 kg/m2; Mallampatti class: III-IV; Reduced mouth opening < 4 cm; Neck circumference > 40 cm for females and > 43 cm for males; Thyromental distance < 6 cm; Ratio of the patient's height to thyromental distance ≥ 23.5; Sternomental distance < 12 cm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- McGrath Mac intubations (Experimental): All 100 patients will be intubated using the McGRATH® MAC video laryngoscope, either through direct or indirect vision laryngoscopy. The liquid crystal display (LCD) monitor of the McGRATH™ MAC was initially covered; if the anesthesiologist visualized a modified C-L grade 1-3 view, the patient was intubated utilizing this direct view. If the anesthesiologist observed a modified C-L grade 4 view during their initial direct view, the patient was intubated using the indirect method. If intubation via direct laryngoscopy was unsuccessful on the first attempt, the patient was intubated using the indirect view. If both methods of laryngoscopy were unsuccessful, the rescue intubation technique was performed at the discretion of the anesthesiologist.
  Interventions: Device: McGrath MAC enhanced direct laryngoscope

INTERVENTIONS:
Device: McGrath MAC enhanced direct laryngoscope — The McGRATH® MAC enhanced direct laryngoscope (EDL) combines the familiarity of direct laryngoscopy with an inline video camera for an enhanced view.
  All 100 patients will be intubated using the McGRATH® MAC video laryngoscope, either through direct or indirect vision laryngoscopy. The LCD monitor of the McGRATH™ MAC was initially covered; if the anesthesiologist visualized a modified C-L grade 1-3 view, the patient was intubated utilizing this direct view. If the anesthesiologist observed a modified C-L grade 4 view during their initial direct view, the patient was intubated using the indirect method. If intubation via direct laryngoscopy was unsuccessful on the first attempt, the patient was intubated using the indirect view. If both methods of laryngoscopy were unsuccessful, the rescue intubation technique was performed at the discretion of the anesthesiologist.

SUMMARY:
This study was designed to determine the first attempt success rate of tracheal intubation with the McGRATH™ MAC laryngoscope using direct visualization in patients with known difficult airways, as well as exploring the possibility of identifying a particular direct Cormack-Lehane (C-L) grade view where indirect (video) visualization can be most beneficial during laryngoscopy and intubation.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 50 kg/m2
* Two or more of the following inclusion criteria: Mallampati class: III-IV; Reduced mouth opening < 4 cm; Neck circumference > 40 cm for females and > 43 cm for males; Thyromental distance < 6 cm; Ratio of the patient's height to thyromental distance ≥ 23.5; Sternomental distance < 12 cm

Exclusion Criteria:

* BMI ≥ 50 kg/m2
* emergency status
* cervical injury or pathology
* neck irradiation
* known difficult airway
* risk of gastric aspiration
* hemodynamic instability
* requiring rapid sequence intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carin A Hagberg, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Device information — http://www.medtronic.com/covidien/en-us/products/intubation/mcgrath-mac-video-laryngoscope.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | McGrath Mac Intubations
Started | 100
Completed | 99
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- McGrath Mac Intubations: All 100 patients will be intubated using the McGRATH® MAC video laryngoscope, either through direct or indirect vision laryngoscopy. The LCD monitor of the McGRATH™ MAC was initially covered; if the anesthesiologist visualized a modified C-L grade 1-3 view, the patient was intubated utilizing this direct view. If the anesthesiologist observed a modified C-L grade 4 view during their initial direct view, the patient was intubated using the indirect method. If intubation via direct laryngoscopy was unsuccessful on the first attempt, the patient was intubated using the indirect view. If both methods of laryngoscopy were unsuccessful, the rescue intubation technique was performed at the discretion of the anesthesiologist.
Arm/Group | McGrath Mac Intubations
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] — Age is reported not for 100 subjects, but only for the 94 who were analyzed. Of the 100 patients recruited, 6 patients were excluded from data analysis. 4 patients were found to not meet inclusion criteria. One patient with glottic view grade 3 was erroneously intubated via the indirect method. For another patient, the anesthesiologist aborted the protocol due to encountered difficulties. Population: Of the 100 patients recruited, 6 patients were excluded from data analysis. 4 patients were found to not meet inclusion criteria. One patient with glottic view grade 3 was erroneously intubated via the indirect method. For another patient, the anesthesiologist aborted the protocol due to encountered difficulties.
  years
    number analyzed (Participants) | 94
    (all) | 53.17 (14.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Successfully Intubated on First Attempt With Use of Either a Direct or Indirect Laryngoscopic View
Description: All 100 patients will be intubated using the McGRATH® MAC video laryngoscope, either through direct or indirect vision laryngoscopy. The LCD monitor of the McGRATH™ MAC was initially covered; if the anesthesiologist visualized a modified C-L grade 1-3 view, the patient was intubated utilizing this direct view. If the anesthesiologist observed a modified C-L grade 4 view during their initial direct view, the patient was intubated using the indirect method. If intubation via direct laryngoscopy was unsuccessful on the first attempt, the patient was intubated using the indirect view. If both methods of laryngoscopy were unsuccessful, the rescue intubation technique was performed at the discretion of the anesthesiologist.
Time Frame: after successful endotracheal tube placement
Population: Of the 100 patients recruited, 6 patients were excluded from data analysis. 4 patients were found to not meet inclusion criteria. One patient with glottic view grade 3 was erroneously intubated via the indirect method. For another patient, the anesthesiologist aborted the protocol due to encountered difficulties.
Measure: Count of Participants; unit: Participants
Arm/Group | McGrath Mac Intubations
Number analyzed (Participants) | 94
Participants
  direct laryngoscopic view | 72
  indirect laryngoscopic view | 16

2. Secondary Outcome: Glottic View With Direct Laryngoscopy
Description: Glottic view as described by Cormack and Lehane, scored as follows- Grade 1. Full view of glottis Grade 2a. Partial view of glottis Grade 2b. Arytenoids or posterior portion of cords just visible Grade 3. Only the epiglottis visible Grade 4. Neither epiglottis nor glottis visible
Time Frame: at the time of laryngoscopy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | McGrath Mac Intubations
Number analyzed (Participants) | 94
Participants
  Grade 1 view | 11
  Grade 2a view | 18
  Grade 2b view | 27
  Grade 3 view | 21
  Grade 4 view | 17

3. Secondary Outcome: Glottic View With Indirect Laryngoscopy
Description: Glottic view as described by Cormack and Lehane (Samsoon GL, Young JR. Difficult tracheal intubation: A retrospective study. Anesthesia 1987; 42:487), scored as follows- Grade 1. Full view of glottis Grade 2a. Partial view of glottis Grade 2b. Arytenoids or posterior portion of cords just visible Grade 3. Only the epiglottis visible Grade 4. Neither epiglottis nor glottis visible
Time Frame: at the time of laryngoscopy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | McGrath Mac Intubations
Number analyzed (Participants) | 94
Participants
  Grade 1 view | 51
  Grade 2b view | 17
  Grade 2a view | 16
  Grade 3 view | 6
  Grade 4 view | 4

4. Secondary Outcome: Time for Direct View Laryngoscopy During the First Attempt
Description: Time from mouth opening to best direct laryngoscopic view
Time Frame: at the time of laryngoscopy
Population: Of the 100 patients recruited, 6 patients were excluded from data analysis, as describe in Outcome Measure 1's Analysis Population Description. 78 of the 94 analyzed had direct laryngoscopy, and thus 78 are analyzed in this outcome measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | McGrath Mac Intubations
Number analyzed (Participants) | 78
seconds | 12.41 (7.13)

5. Secondary Outcome: Time for Indirect View Laryngoscopy During the First Attempt
Description: Time from mouth opening to best indirect laryngoscopic view
Time Frame: at the time of laryngoscopy
Population: Of the 100 patients recruited, 6 patients were excluded from data analysis, as describe in Outcome Measure 1's Analysis Population Description. 16 of the 94 analyzed had direct laryngoscopy, and thus 16 are analyzed in this outcome measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | McGrath Mac Intubations
Number analyzed (Participants) | 16
seconds | 14.73 (9.99)

6. Secondary Outcome: Time for Intubation
Description: Time for laryngoscopy (either direct or indirect) plus the time for endotracheal tube (ETT) cuff to pass vocal cords.
Time Frame: at the time of laryngoscopy
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | McGrath Mac Intubations
Number analyzed (Participants) | 94
seconds | 35.91 (22.66)

7. Secondary Outcome: Number of Intubation Attempts
Time Frame: at the time of intubation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | McGrath Mac Intubations
Number analyzed (Participants) | 94
Participants
  1 attempt | 88
  2 attempts | 5
  3 attempts | 1

8. Secondary Outcome: Number of Participants Who Received External Laryngeal Manipulation During the First Attempt
Time Frame: at the time of intubation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | McGrath Mac Intubations
Number analyzed (Participants) | 94
Participants | 42

9. Secondary Outcome: Number of Participants on Whom Bougie (Introducer) Was Used to Facilitate Intubation on the First Attempt
Time Frame: at the time of intubation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | McGrath Mac Intubations
Number analyzed (Participants) | 94
Participants | 12

10. Secondary Outcome: Subjective Ease of Laryngoscopy
Description: The anesthesiologists rated the McGRATH™ MAC's ability in managing airways as "very easy," "easy," "slight resistance," "difficult," or "not possible." The difficulty of laryngoscopy was evaluated during the insertion and placement of the McGRATH™ MAC, from the patient's lips, into their oropharynx, until a glottic view was obtained.
Time Frame: at the time of laryngoscopy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | McGrath Mac Intubations
Number analyzed (Participants) | 94
Participants
  very easy | 22
  easy | 29
  slight resistance | 23
  difficult | 19
  not possible | 1

11. Secondary Outcome: Subjective Ease of Intubation
Description: The anesthesiologists rated the McGRATH™ MAC's ability in managing airways as "very easy," "easy," "slight resistance," "difficult," or "not possible." The difficulty of endotracheal tube (ETT) delivery (that is, intubation) was evaluated during the insertion of the ETT into the patient's mouth, until the ETT passed the vocal cords.
Time Frame: at the time of laryngoscopy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | McGrath Mac Intubations
Number analyzed (Participants) | 94
Participants
  very easy | 20
  easy | 39
  slight resistance | 21
  difficult | 13
  not possible | 1

ADVERSE EVENTS:
Time Frame: Adverse Event data include measures of post-operative discomfort upon entering the Post-Anesthesia Care Unit (PACU). Patients enter the PACU within 30 minutes of completion of surgery, and they leave the PACU approximately 1-2 hours after entering the PACU.
Description: All 100 patients were assessed for SAEs. 94 patients were assessed for other AEs (not including SAEs): 6 patients were excluded from data analysis; 4 patients were found to not meet inclusion criteria; one patient with glottic view grade 3 was erroneously intubated via the indirect method; and for another patient, the anesthesiologist aborted the protocol due to encountered difficulties.
Arm/Group | McGrath Mac Intubations
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 48/94
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | McGrath Mac Intubations (N=94)
Hoarseness (General disorders) | 41 (41)
Sore mouth (General disorders) | 8 (8)
sore neck (General disorders) | 7 (7)
Sore jaw (General disorders) | 2 (2)
Dysphonia (General disorders) | 4 (4)
Dysphagia (General disorders) | 10 (10)
Alteration in Tongue (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes